CLINICAL TRIAL: NCT07133607
Title: Effectiveness of a Pain Neuroscience Education and Therapeutic Exercise Program Delivered by Primary Care Physiotherapists to Patients With Chronic Nociplastic Spinal Pain: a Multicenter Randomized Controlled Trial.
Brief Title: Effectiveness of a Pain Neuroscience Education and Therapeutic Exercise Program Delivered by Primary Care Physiotherapists to Patients With Chronic Nociplastic Spinal Pain
Acronym: AP-AADC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Distrito de Atención Primaria Sevilla (Other)
Collaborators: Junta de Andalucia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FISIOTERAPIA3; AP-AADC (Other: Health Department of the Andalusian Regional Government)
Record Dates: First submitted 2025-07-22; First posted 2025-08-21 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain (Back / Neck)
Keywords: pain chronic; central sensibilitation; public health system; pain education; physiotherapy; somatosensory; body outline; therapeutic physical exercise
MeSH Terms: conditions — Chronic Pain | interventions — Exercise; Hyperthermia, Induced

STUDY DESIGN:
Intervention Model Description: parallel study for three interventions groups
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Active Comparator): The patients will receive the usual physiotherapy treatment provided in Primary Care Physiotherapy units, supported by the current Primary Care Physiotherapy protocols of Castilla y León (33), since Andalusia does not currently have any published. The patient will receive 12 sessions of thermotherapy (Infrared/Microwave) and analgesic electrotherapy (analgesic Tens currents) in the painful area(s), and will be prescribed exercises recommended by the Spanish Society of Physical Medicine and Rehabilitation (SERMEF) (34). The learning and execution of the exercises will be supervised by a Primary Care physiotherapist. The sessions will be with a frequency of 2 per week on alternate days for 6 weeks.
  Interventions: Other: Classic physiotherapy treatment with physical exercise, analgesic electrotherapy and thermotherapy
- intervention type 1, education to pain and physical exercise (Experimental): The sessions will be conducted in groups of 10 to 15 patients.
  * 4 pain science education sessions, each lasting 1.5 hours (6 hours), with one session per week, for 4 weeks.
  * 12 therapeutic physical exercise program sessions, each lasting 1 hour, to be conducted over 6 weeks (12 hours), with two sessions per week. Although the intervention is group-based, individual instructions will be given to patients. Reference will be made to the content learned in the neuroeducation sessions. The exercise dose must be adjusted to the patient's condition, keeping in mind that, due to the inhibition of the descending pain modulation system, they may experience an initial increase in pain during the first sessions, so as not to alarm the patient and prevent the activity from being discontinued. The main objective is to increase the patient's functionality, an aspect that will be constantly reinforced.
  The session structure will be as recommended by the American College of Sports Medicine, with se
  Interventions: Other: education about pain and physical excersice
- intervention type 2, education to pain and physical exercise with somatosensorial treatment (Experimental): Patients assigned to this group will receive, in addition to the same intervention as the AADC study group "intervention type 2", somatosensory and body schema treatment for the changes observed in an initial assessment during the 4 weeks prior.
  The prescribed treatment will be repeated daily at home. To facilitate
  the progress of the treatment, it is recommended that a companion participate in the first session, when possible, where the daily intervention to be performed at home will be explained.
  If the participation of a companion is not possible, the patient will attend the Health Center's physiotherapy room once a day to be accompanied by the physiotherapist and offered the same treatment opportunities.
  As a control and monitoring measure, the patient will attend the physiotherapy room once a week and will be called again weekly to verify that the treatment is being performed correctly. They will also be provided with a form to record their home treatment.
  Interventions: Other: education about pain and physical excersice with somatosensorial treatment

INTERVENTIONS:
Other: education about pain and physical excersice — The sessions will be conducted in groups of 10 to 15 patients.
  * 4 pain science education sessions, each lasting 1.5 hours (6 hours), with one session per week, for 4 weeks.
  * 12 therapeutic physical exercise program sessions, each lasting 1 hour, to be conducted over 6 weeks (12 hours), with two sessions per week. Although the intervention is group-based, individual instructions will be given to patients. Reference will be made to the content learned in the neuroeducation sessions. The exercise dose must be adjusted to the patient's condition, keeping in mind that, due to the inhibition of the descending pain modulation system, they may experience an initial increase in pain during the first sessions, so as not to alarm the patient and prevent the activity from being discontinued. The main objective is to increase the patient's functionality, an aspect that will be constantly reinforced.
  The session structure will be as recommended by the American College of Sports Medicine, with se
  Arms: intervention type 1, education to pain and physical exercise
Other: education about pain and physical excersice with somatosensorial treatment — Patients assigned to this group will receive, in addition to the same intervention as the AADC study group "intervention type 2" (education about pain), somatosensory and body schema treatment for the changes observed in an initial assessment during the 4 weeks prior.
  The prescribed treatment will be repeated daily at home. To facilitate
  the progress of the treatment, it is recommended that a companion participate in the first session, when possible, where the daily intervention to be performed at home will be explained.
  If the participation of a companion is not possible, the patient will attend the Health Center's physiotherapy room once a day to be accompanied by the physiotherapist and offered the same treatment opportunities.
  As a control and monitoring measure, the patient will attend the physiotherapy room once a week and will be called again weekly to verify that the treatment is being performed correctly. They will also be provided with a form to record their home treatment.
  Arms: intervention type 2, education to pain and physical exercise with somatosensorial treatment
Other: Classic physiotherapy treatment with physical exercise, analgesic electrotherapy and thermotherapy — The patients will receive the usual physiotherapy treatment provided in Primary Care Physiotherapy units, supported by the current Primary Care Physiotherapy protocols of Castilla y León, since Andalusia does not currently have any published. The patient will receive 12 sessions of thermotherapy (Infrared/Microwave) and analgesic electrotherapy (analgesic Tens currents) in the painful area(s), and will be prescribed exercises recommended by the Spanish Society of Physical Medicine and Rehabilitation (SERMEF). The learning and execution of the exercises will be supervised by a Primary Care physiotherapist. The sessions will be with a frequency of 2 per week on alternate days for 6 weeks.
  Arms: control group

SUMMARY:
The main objective of the project is to evaluate the effectiveness, in terms of quality of life, of a therapy based on an Active Coping Protocol for Non-Cancer Chronic Pain in the Primary Care setting. This approach involves no medications or invasive procedures and is based on pain neuroscience education and physical exercise, either alone or combined with treatment targeting body schema and somatosensory disturbances. The comparison will be made against a treatment involving thermotherapy and traditional physical exercise.

One of the most well-documented national primary care experiences combining pain neuroeducation and physical exercise, with a detailed methodology, was carried out by the Health System of Castilla y León (Sacyl) in Valladolid. It yielded significant results using a protocol consisting of 6 sessions of pain neuroscience education and 18 sessions of group exercise.

Based on this reference study, two hypotheses are proposed: the first is that reducing the number of sessions in the Active Coping Protocol for Chronic Pain would maintain treatment effectiveness. The second hypothesis suggests the potential for improved outcomes by combining the Active Coping Protocol with body schema and somatosensory disturbance treatment.

To test these hypotheses, a randomized experimental study with three parallel groups will be conducted on patients aged 18 to 70, referred to Physiotherapy from health centers in the Sevilla Health District. These patients experience daily spinal chronic pain for more than 3 months or on at least half of the days over more than 6 months, with central sensitization as the underlying cause.

Effectiveness will be measured in terms of quality of life (SF-36), pain intensity (Visual Analog Scale), satisfaction level, kinesiophobia, catastrophizing, pressure pain threshold, disability index (NDI/Oswestry), medication reduction, and number of monthly medical appointments.

Secondary objectives include evaluating, in both experimental groups compared to the control, the outcome variables: pain intensity, treatment adherence, kinesiophobia, catastrophizing, pressure pain threshold, descending modulation system, lumbar disability index, severity level, anxiety, sleep quality, analgesic consumption, healthcare visits, and satisfaction with care received.

A sample size of 135 patients has been calculated and will be randomized into the three study groups. The control group will receive thermotherapy-electrotherapy and conventional therapeutic exercise. Experimental group 1 will follow the Active Coping Program for Chronic Pain (4 education sessions and 12 physical exercise sessions). Experimental group 2 will receive somatosensory and body schema treatment along with the Active Coping Program.

The study is evaluator-blinded. Statistical analysis will be performed using SPSS version 28 and R Core Team (2023). Statistical significance will be set at p-values <0.05. Authorization will be requested from the relevant Research Ethics Committee.

The results of this study may lead to updates of existing protocols, development of guidelines and manuals for managing chronic musculoskeletal pain, ongoing training for primary care professionals, and publication in high-impact scientific journals to disseminate knowledge.

ELIGIBILITY:
Inclusion Criteria:

* Users of the Public Health System of Andalusia, registered in the User Database (BDU) of the Sevilla Health District.
* Ages between 18 and 70.
* Chronic lumbar pain lasting more than 3 months, likely due to central sensitization (likely nociplastic pain).
* The diagnosis of Central Sensitization will be made according to the most recent algorithm published by Nijs et al. in Lancet.

Exclusion Criteria:

* Oncological pain (pain related to cancer)
* Spinal fracture or spinal surgery in the previous year.
* Neurological cognitive impairment that prevents understanding of pain neuroeducation (if in doubt, the Minimental Test will be performed, requiring a minimum score of 25)
* Physical conditioning deficit that prevents the execution of the Physical --Education program (minimum requirement: normal execution time of <10 seconds for the timed "Up and Go" test).
* Pregnancy
* Cauda equina syndrome
* Chronic fatigue syndrome
* Fibromyalgia
* Complex Regional Pain Syndrome
* Clinical conditions that may aggravate chronic spinal pain.
* Associated pathologies that prevent the performance of a physical exercise program (myopathies and neurological disorders).
* Currently undergoing alternative therapies.
* The presence of pain in other anatomical regions, apart from spinal pain, is not a reason for exclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the value of quality of life measured Trough sf 36 questionnaire at 6 Months | from the start of treatment, at 11 weeks and at 26 weeks
  0 equals very poor quality of life and 100 very good quality of life

SECONDARY OUTCOMES:
Change from Baseline in the value of pain intensitivity measured trough AVS scale at 6 Months | from the start of treatment, at 11 weeks and at 26 weeks
  0 equals absence of pain and 10 a lot of pain
Change from Baseline in the value of regular physical activity measured Trough international physical activity questionnaire (IPAQ)at 6 Months | from the start of treatment, at 11 weeks and at 26 weeks
  low/moderate/high
Change from Baseline in the value of kinesophobia measured Trough kinesophobia questionnaireTampa-TSK-11SV at 6 Months | from the start of treatment, at 11 weeks and at 26 weeks
  The lowest possible score, 11, denotes negligible or nonexistent kinesiophobia. The highest possible score, 44, denotes a severe fear of experiencing pain when moving.
Change from Baseline in the value of Pain Catastrophizing measured Trough Pain Catastrophizing Scale (PCS) at 6 Months | from the start of treatment, at 11 weeks and at 26 weeks
  Together with three subscale scores assessing rumination, magnification, and helplessness, the overall score has a range of 0-52.
  Higher scores indicate a greater degree of pain catastrophizing. A total score >30 represents a clinically significant level of pain catastrophizing.
Change from Baseline in the value of pain threshold to pressure at 6 Months trough the protocol described in the study by Neziri et al, measuring four points using the procedure described by Fisher | from the start of treatment, at 11 weeks and at 26 weeks
  A pain threshold below 4 kg/cm2 identifies increased sensitivity to pressure.
Change from Baseline in the value of Conditional pain modulation system at 6 Months trough Protocol validated by Larsen et al. | from the start of treatment, at 11 weeks and at 26 weeks
  The UDP is assessed in the anterior tibial muscle (three times to calculate the mean), then, using a conditioning clamp, a tonic pain stimulus is applied by pinching the earlobe for 60 seconds (10). When the VAS of earlobe pain exceeds 60 mm, the pressure pain threshold in the anterior tibial muscle is assessed again three times. The CPM effect is calculated as the percentage change [(conditioning/baseline × 100) - 100] and the difference [conditioning-baseline] in the pressure pain threshold as recommended by Yamitsky D. et al.
Change from Baseline in the value of lumbar disability index measured Trough Rolland Morris Scale at 6 Months | from the start of treatment, at 11 weeks and at 26 weeks
  The final score, out of 24 represents the degree of disability due to low back pain. A maximum score of 24 indicates the greatest degree of disability from back pain.
Change from Baseline in the value of Level of severity of the case at 6 Months trough the Central Sensitization Inventory | from the start of treatment, at 11 weeks and at 26 weeks
  0 equals absence of severity associated with central sensitization and 100 a lot of severity associated
Change from Baseline in the value of sleep quality and patterns in adults of the case at 6 Months trough The Pittsburgh Sleep Quality Questionnaire (PSQI) | from the start of treatment, at 11 weeks and at 26 weeks
  It provides a global measure of sleep quality, with a range of 0 to 21, where scores greater than 5 suggest significant alterations in sleep quality
Change from Baseline in the value of Medication intake of the case at 6 Months trough a survey | from the start of treatment, at 11 weeks and at 26 weeks
  The results will be expressed in weekly doses according to the type of drug taken.
During the follow-up period, visits to the family doctor, emergency services, and specialists will be recorded using the Digital Health Record. | from the start of treatment, at 11 weeks and at 26 weeks
Change from Baseline in the value of satisfaction with health services of the case at 6 Months trough The Spanish version of the Client Satisfaction Questionnaire (CSQ-8) | from the start of treatment, at 11 weeks and at 26 weeks
Change from Baseline in the value of Regular physical activity of the case at 6 Months trough International Physical Activity Questionnaire (IPAQ). | from the start of treatment, at 11 weeks and at 26 weeks
Change from Baseline in the value of fatigue intensitivity measured trough AVS scale at 6 Months | from the start of treatment, at 11 weeks and at 26 weeks
  0 equals absence of fatigue and 10 a lot of fatigue
Change from Baseline in the value of short stress test at 6 Months trough number of squats in 30 seconds, 60 seconds, and modified Borg scale of perceived exertion | from the start of treatment, at 11 weeks and at 26 weeks
  0 equals absence of perceived exertion and 10 a lot of perceived exertion
Change from Baseline in the value of Flamingo Balance Test at 6 Months trough number of times you need to land in 30" | from the start of treatment, at 11 weeks and at 26 weeks

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galan-Martin MA, Montero-Cuadrado F, Lluch-Girbes E, Coca-Lopez MC, Mayo-Iscar A, Cuesta-Vargas A. Pain neuroscience education and physical exercise for patients with chronic spinal pain in primary healthcare: a randomised trial protocol. BMC Musculoskelet Disord. 2019 Nov 3;20(1):505. doi: 10.1186/s12891-019-2889-1. PMID 31679512